CLINICAL TRIAL: NCT02966249
Title: Comparison of Dexmetomidine's Efficacy as an Adjuvant to Intrathecal Levobupivacaine and Intravenous Administration Additionally to Spinal Anaesthesia, In Total Knee Arthroplasty
Brief Title: Dexmetomidine Intrathecally and Intravenously Additionally to Spinal Anaesthesia, in Total Knee Arthroplasty
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: KAT General Hospital (Other)
Responsible Party: Principal Investigator, Ioanna Diagoupi, Intern doctor in anaesthesiology, KAT General Hospital
Allocation: Randomized | Model: Factorial | Masking: Double | Purpose: Treatment
Other Study IDs: 9092
Record Dates: First submitted 2016-08-28; First posted 2016-11-17 (Estimated); Last update posted 2016-11-17 (Estimated); Status verified 2016-10

CONDITIONS: Neuromuscular Block
Keywords: dexmetomidine, intrathecally, intavenously,anesthesia
MeSH Terms: interventions — Levobupivacaine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (6):
- Levobupivacaine intrathecally (Other): 3 ml Levobupivacaine 0,5% (15mg) given intrathecally once for anesthesia in total knee arthroplasty
  Interventions: Drug: Levobupivacaine; Drug: Normal Saline intrathecally
- Dexmetomidine intrathecally (Active Comparator): 5 μgr Dexmetomidine given intrathecally once for anesthesia in total knee arthroplasty
  Interventions: Drug: Levobupivacaine; Drug: Normal Saline added intrathecally; Drug: Dexmetomidine intrathecally
- Dexmetomidine intravenously (Active Comparator): Continuous infusion of dexdemetomidine at a rate of 0.25 μg/kg/h given intravenously starting 10 min before spinal anesthesia in total knee arthroplasty
  Interventions: Drug: Levobupivacaine; Drug: Dexmetomidine intravenously; Drug: Ringer's Lactate solution intravenously
- Normal Saline intrathecally (Placebo Comparator): 0,5 ml Normal Saline given intrathecally given once for spinal anesthesia in total knee arthroplasty
  Interventions: Drug: Levobupivacaine; Drug: Normal Saline added intrathecally; Drug: Dexmetomidine intrathecally
- Normal Saline added intrathecally (Other): Normal Saline added intrathecally up to 0,5 ml given intrathecally for spinal anesthesia in total knee arthroplasty
  Interventions: Drug: Levobupivacaine; Drug: Normal Saline intrathecally; Drug: Dexmetomidine intrathecally
- Ringer's Lactate solution intravenously (Other): Continuous infusion of Ringer's Lactate solution given intravenously for total knee arthroplasty will start 10 minutes before spinal anesthesia to the end of the operation
  Interventions: Drug: Levobupivacaine; Drug: Dexmetomidine intravenously; Drug: Ringer's Lactate solution intravenously

INTERVENTIONS:
Drug: Levobupivacaine — 3 ml Levobupivacaine 0.5% (15mg) given intrathecally
  Other Names: LB
Drug: Dexmetomidine intravenously — Continuous infusion of dexdemetomidine at a rate of 0.25 μg/kg/h given intravenously 10 min before spinal anesthesia in total knee arthroplasty
  Other Names: DEX
  Arms: Dexmetomidine intravenously; Ringer's Lactate solution intravenously
Drug: Normal Saline added intrathecally — Normal Saline added to 5μgr dexmetomidine up to 0,5 ml given intrathecally for spinal anesthesia in total knee arthroplasty
  Other Names: N/S
  Arms: Dexmetomidine intrathecally; Normal Saline intrathecally
Drug: Normal Saline intrathecally — 0,5 ml Normal Saline given intrathecally given once for spinal anesthesia in total knee arthroplasty
  Other Names: N/S
  Arms: Levobupivacaine intrathecally; Normal Saline added intrathecally
Drug: Ringer's Lactate solution intravenously — Continuous infusion of Ringer's Lactate solution given intravenously, starting 10 minutes before spinal anesthesia up to the end of the operation
  Other Names: R/L
  Arms: Dexmetomidine intravenously; Ringer's Lactate solution intravenously
Drug: Dexmetomidine intrathecally — 5 μgr dexmetomidine given intrathecally once for anesthesia in total knee replacement
  Other Names: DEX
  Arms: Dexmetomidine intrathecally; Normal Saline added intrathecally; Normal Saline intrathecally

SUMMARY:
The present study is designed to evaluate and compare the efficacy of intrathecal dexmedetomidine (DEX) as an adjuvant to Levobupivacaine in spinal anaesthesia and DEX's intravenous administration, without loading dose, additionally to spinal anaesthesia, in patients undergoing total knee arthroplasty.

DETAILED DESCRIPTION:
Introduction

Various adjuvants like morphine, fentanyl, clonidine, ketamine are being used since long for improvement of intraoperative anaesthesia and postoperative analgesia following spinal anaesthesia. On the other hand, such adjuvants have their associated adverse effects. As a result, search for an effective adjuvant is still going on. Dexmedetomidine (DEX), a selective α2-adrenoceptor agonist, has analgesic and sedative effects and nowadays, is being studied for its adjuvant action in subarachnoid anaesthesia.

As far as DEX is concerned, it has been reported that it can be administered intravenously in additional to spinal anaesthesia, in order to promote sensory and motor blockade duration and postoperative analgesia, because of its synergistic action with local anaesthetics.

DEX is a highly selective alpha 2 adrenergic receptor agonist with a higher α2/α1 selectivity ratio of 1620:1 than clonidine (200:1). It was first introduced to clinical as a sedative in intensive care unit. Alpha-2 adrenergic receptor agonists have been tried by many clinicians due to their sedative, anxiolytic, hypnotic, analgesic, perioperative sympatholytic and stable haemodynamic properties. DEX, specifically, has all these properties, without causing respiratory depression. Currently its adjuvant action in spinal anaesthesia and its intravenous administration, additionally to subarachnoid anaesthesia, is being explored.

Aim The present study is designed to evaluate and compare the efficacy of intrathecal DEX as an adjuvant to Levobupivacaine in spinal anaesthesia and DEX's intravenous administration, without loading dose, additionally to spinal anaesthesia, in patients undergoing total knee arthroplasty.

Material and Methods It will be a prospective, double blind study among 90 adult patients, undergoing total knee arthroplasty under spinal anaesthesia. This study has been approved by the Institutional Medical Ethics Committee of KAT Hospital of Athens City. Informed consent will be obtained from all subjects.

The patients will be randomly allocated to 3 groups (Group I, Group II, and Group III) of 30 each. Group I will receive 3 ml Levobupivacaine 0,5 % ( 15 mg ) and normal saline intrathecally. Group II will receive Levobupivacaine 0,5% and DEX (5 μg) made up to 0,5 ml with normal saline intrathecally. Group III will receive Levobupivacaine 0,5% and normal saline and DEX in Ringer Solution intravenous at a rate of 0.25 μg/kg/h. Intravenous infusion will start 10 minutes before spinal anesthesia and will last until the end of the operation.

The onset and duration of sensory and motor block, the duration of postoperative analgesia, hemodynamic parameters intraoperatively and postoperatively and adverse effects will be recorded.

Hemodynamic parameters such as arterial pressure and blood pulse will be recorded every 5 minutes for the first 30 minutes, thereafter every 10 minutes till the end of surgery.

Sedation scores will be assessed every 15 minutes intraoperatively using the Ramsay Sedation Scale, which is :

If Awake

* Ramsey 1 Anxious, agitated, restless
* Ramsey 2 Cooperative, oriented, tranquil
* Ramsey 3 Responsive to commands only If Asleep
* Ramsey 4 Brisk response to light glabellar tap or loud auditory stimulus
* Ramsey 5 Sluggish response to light glabellar tap or loud auditory stimulus
* Ramsey 6 No response to light glabellar tap or loud auditory stimulus Side effects like sedation, nausea, vomiting, shivering will be recorded intraoperatively and postoperatively.

ELIGIBILITY:
Inclusion Criteria:

* Patients selected for total knee arthroplasty of approximately one and half hour (90 min) duration under spinal anaesthesia.
* Patients who belong to American Society of Anaesthesiologists (ASA) physical status grade I and II

Exclusion Criteria:• Patients with coagulation and neurological disorders

* Patients allergic to DEX
* Patients showing unwillingness for spinal anaesthesia

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2016-10; Primary Completion 2017-04 (Estimated); Study Completion 2017-09 (Estimated)

PRIMARY OUTCOMES:
Onset and duration of sensory block using the ' pin-prick ' method,in total knee athroplasty, using DEX as an adjuvant to intrathecal Levobuvicaine and iv administration additionally to spinal anesthesia with Levobuvicaine | The time of onset will be taken from the time of injection of drug intrathecally to loss of pinprick sensation to T12 within 30 min. Duration of sensory blockade will be measured as time from onset to time of return of piniprick sensation to S1 level.
  By using a hypodermic needle at 2 min interval, we will assess the 'pin-prick' sensation from T12 to S1 The onset of sensory block will be tested by 'pin-prick method' using a hypodermic needle at 2 minutes interval. The time of onset will be taken from the time of injection of drug into subarachnoid space to loss of pinprick sensation to T12 level. We study 90 patients(ASAI-II) devided in 3 groups and we measure the highest level of sensory block, time for two dermatomal segments regression of sensory level, duration of sensory blockade taken as time from onset to time of return of pinprick sensation to S1 (heel) dermatomal area will be noted.
Onset and duration of motor block using the Modified Bromage Scale, in total knee athroplasty, using DEX as an adjuvant to intrathecal Levobuvicaine and iv administration additionally to spinal anesthesia with Levobuvicaine | Onset time will be taken from the time of injection of drug intrathecally to the patient's inability to lift the extended leg within 30 min. The duration will be taken from time of injection of drug to the patient's ability to lift the extended leg.
  By using the Modified Bromage Scale we will assess the onset and duration of motor block. Grade 0 : Full flexion of knees and feet. Grade 1: Just able to flex knees, full flexion of feet. Grade 2: Unable to flex knees, but some flexion of feet possible. Grade 3; Unable to move legs or feet.
Duration of post-operative analgesia using the Visual Analogue Scale (VAS), in total knee arthroplasty, using DEX as an adjuvant to intrathecal Levobuvicaine and iv administration additionally to spinal anesthesia with Levobuvicaine | We will record the post-operative analgesia using the Visual Analogue Scale (VAS) at the end of the surgery and 3, 6, 12,24 hours after the end of the surgeryn and at the end of the surgery. an interval of 3, 6 ,and 12 h after surgery
  VAS is a scale from 0 to 10, with 0 indicating 'no pain' and 10 indicating the most severe pain, that somebody has experienced. Rescue analgesics will be given to the patients when VAS>3, which will be the cut-off point of our study.

SECONDARY OUTCOMES:
Hemodynamic stability of DEX, used as an adjuvant to intrathecal Levobupivacaine and intravenous administration additionally to spinal anesthesia, in total knee arthroplasy | SAP will be recorded at the time of the spinal injection, 10, 20, 30,45, 60 min after spinal injection and at the end of the surgery.
  We will record SAP intra-operatively
Hemodynamic stability of DEX, used as an adjuvant to intrathecal Levobupivacaine and intravenous administration additionally to spinal anesthesia, in total knee arthroplasy | DAP will be recorded will be recorded at the time of the spinal injection, 10, 20, 30,45, 60 min after spinal injection and at the end of the surgery.
  We will record DAP intra-operatively
Hemodynamic stability of DEX, used as an adjuvant to intrathecal Levobupivacaine and intravenous administration additionally to spinal anesthesia, in total knee arthroplasy | HR will be recorded will be recorded at the time of the spinal injection, 10, 20, 30,45, 60 min after spinal injection and at the end of the surgery.
  We will record HR intra-operatively
Adverse effects of DEX, used as an adjuvant to intrathecal Levobupivacaine and intravenous administration additionally to spinal anaesthesia with Levobupivacaine, in total knee arthroplasy | Adverse effects will be recorded will be recorded at the time of the spinal injection, 15, 30, 60 min after spinal injection, at the end of the surgery and 3, 6, 12, 24 hours after the end of the surgery
  We will record adverse effects like nausea, vomitting and shivering.
Sedation will be assessed with the Ramsay Sedation Scale, in total knee arthroplasty, by using DEX as an adjuvant to intrathecal Levobupivacaine and intravenous administration additionally to spinal anesthesia with Levobuvicaine | Sedation scores will be assessed will be recorded at the time of the spinal injection, 10, 20, 30,45, 60 min after spinal injection, at the end of the surgery and 30 minutes after the end of the surgery
  The Ramay Sedation Scale is : If awake : Ramsay 1 Anxious, agitated, restless Ramsay 2 Co-operative, oriented,tranquil, Ramsay 3 Responsive to commands only. If asleep: Ramsey 4 Brisk response to light glabellar tap or loud auditory stimulus Ramsey 5 Sluggish response to light glabellar tap or loud auditory stimulus Ramsey 6 No response to light glabellar tap or loud auditory stimulus

CONTACTS AND LOCATIONS:
Overall Officials: Efi Stavropoulou, Study Chair — KAT GENERAL HOSPITAL OF ATTICA; Cathrin Chazapis, Study Chair — KAT General Hospital of Athens
Locations (1):
- Kat General Hospital of Attca, Kifissia, Greece

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Zhang H, Li M, Zhang SY, Fu M, Zhang SY. Intravenous Dexmedetomidine Promotes Spinal Bupivacaine Anesthesia and Postoperative Analgesia in Lower Limb Surgery: A Double-Blind, Randomized Clinical CONSORT Study. Medicine (Baltimore). 2016 Feb;95(8):e2880. doi: 10.1097/MD.0000000000002880. PMID 26937924
- [Background] Chan IA, Maslany JG, Gorman KJ, O'Brien JM, McKay WP. Dexmedetomidine during total knee arthroplasty performed under spinal anesthesia decreases opioid use: a randomized-controlled trial. Can J Anaesth. 2016 May;63(5):569-76. doi: 10.1007/s12630-016-0597-y. Epub 2016 Jan 29. PMID 26830642